CLINICAL TRIAL: NCT00194441
Title: CPP Management Information Feedback and Nursing
Brief Title: Cerebral Perfusion Pressure (CPP) Management Information Feedback and Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Catherine Kirkness, Research Associate Professor,, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14622-C; 5R01NR004901-07 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
Keywords: cerebral circulation; monitoring, physiologic; informatics; nursing care; physiologic variability; outcome; quality adjusted life years
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Highly visible continually updating color coded bar computer display of cerebral perfusion pressure.
  Interventions: Other: Bedside display of cerebral perfusion pressure information
- 2 (Placebo Comparator): Bedside computer display with a blank screen except for a message indicating that the program is running.
  Interventions: Other: Bedside display of cerebral perfusion pressure information

INTERVENTIONS:
Other: Bedside display of cerebral perfusion pressure information — Continually updating highly visible color coded bar graph bedside computer display of cerebral perfusion pressure

SUMMARY:
The aim of the initial proposal was to evaluate, in the context of optimal medical management, the impact of a bedside system of cerebral perfusion pressure (CPP) information feedback on nursing moment-to-moment management of CPP, and the relationship of that management to patient functional outcome at discharge, 3 and 6 months. The primary hypothesis being tested is that Glasgow Outcome Score (GOS) 6 months post acute care discharge will be significantly better in those monitored with the continuous CPP display.

In the second phase of the study the adult study will be extended to children to determine if there is a critical threshold for CPP in children following brain injury based on their outcome at 3, 6, and 12 months. The primary outcome measure is the GOS at 12 months post-injury. The GOS, Behavior Rating Inventory of Executive Function, and PedsQOL will also be assessed at 3, 6, & 12 months, and the Adaptive Behavior Assessment System at 3 and 6 months post-injury. In addition, the researchers will examine variability and complexity of physiologic measures, such as blood pressure, recorded during the intensive care unit stay of adults and children enrolled in the study. The researchers will study the association of these measures with risk for secondary brain injury and ability to predict differences in outcome. The researchers will also assess the value individuals place on varying outcomes following brain injury.

DETAILED DESCRIPTION:
Prevention or reduction of secondary brain injury is a key component in the critical care management of patients with a variety of brain insults. Current clinical management emphasizes maintaining cerebral perfusion pressure (CPP) at or above 70 mm Hg to minimize such secondary brain injury. However, due to poor ergonomics in clinical monitoring displays it is likely that short episodes of decreased CPP are missed by attending nurses in the course of necessary patient repositioning, suctioning, and other routine therapeutic activities. Given the crucial role of neuronal perfusion in preventing secondary injury beyond that of the original brain insult, refining the nurse's ability to visualize and manage CPP on a moment-to-moment basis may allow measurable improvement in short and long-term patient functional outcome. Computer interfaces that provide highly visible information about CPP will be randomly allocated to intensive care unit beds of patients with closed head injury (CHI) or subarachnoid hemorrhage (SAH) in whom intracranial pressure monitors and arterial lines have been placed for medical management, stratified by primary diagnosis (CHI or SAH) and severity. Continuous data will be collected from 150 patients with and 150 patients without the interface monitor for the duration of CPP monitoring. The primary hypothesis being tested is that the Glasgow Outcome Score (GOS) 6 months after acute care discharge will be significantly better in those monitored with the continuous CPP display. Secondary endpoints are GOS at discharge and 3 months after discharge, Functional Independence Measure (FIM) score at discharge, and the Functional Status examination at 3 and 6 months. The percentage of CPP below set levels during hospital monitoring will be determined.

No CPP thresholds have been established that adequately predict how well children who survive a brain injury will do. Thus we will describe the association between various CPP thresholds and children's outcome up to one year after their brain injury. The target number of children to be enrolled is 65.

Studies suggest that the regularity or variability of physiologic measures, for example, heart rate, may give information about how well the system can respond to challenges. Changes in variability may be associated with disease. Describing physiologic variability may therefore be useful to identify critically ill individuals with brain injury who are less able to adapt to challenges and may be a greater risk for further brain injury and poorer outcome.

Measures of the value that individuals place on the various health states are used to calculate quality adjusted life years and assess the cost-effectiveness of treatments. While measures have been developed to assess how individuals value different outcomes, information regarding the value placed on outcomes following brain injury is lacking. We will use these measures to carry out interviews of both brain injury survivors and those who have not had a brain injury to add to the knowledge in this area.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury or subarachnoid hemorrhage
* Age 16 years or older
* Admitted to intensive care unit
* Invasive intracranial pressure and arterial blood pressure monitoring

Exclusion Criteria:

* Impending death

Inclusion Criteria for second phase of study (determination of CPP threshold in children):

* Traumatic brain injury
* Age 15 years or younger
* Able to communicate by telephone
* Admitted to intensive care unit
* Intracranial pressure monitoring

Inclusion Criteria for second phase of study (quality adjusted life years assessment):

* Hospitalized for a traumatic brain injury or subarachnoid hemorrhage at an academic medical center within the last 10 years
* Age 18 years or older at the time of hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1999-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale | Six month follow-up

SECONDARY OUTCOMES:
Glasgow Outcome Scale | Hospital discharge and three month follow-up
Functional Status Examination | Three and six-month follow-up
SF-36 Quality of Life | Six month follow-up
Patient Competency Rating Scale | Six month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Kirkness, PhD, Principal Investigator — University of Washington; Pamela H Mitchell, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Mitchell PH, Burr RL, Kirkness CJ. Information technology and CPP management in neuro intensive care. Acta Neurochir Suppl. 2002;81:163-5. doi: 10.1007/978-3-7091-6738-0_42. PMID 12168293
- [Result] Kirkness CJ, Burr RL, Mitchell PH, Newell DW. Is there a sex difference in the course following traumatic brain injury? Biol Res Nurs. 2004 Apr;5(4):299-310. doi: 10.1177/1099800404263050. PMID 15068659
- [Result] Kirkness CJ, Thompson JM, Ricker BA, Buzaitis A, Newell DW, Dikmen S, Mitchell PH. The impact of aneurysmal subarachnoid hemorrhage on functional outcome. J Neurosci Nurs. 2002 Jun;34(3):134-41. doi: 10.1097/01376517-200206000-00006. PMID 12080869
- [Result] Kirkness CJ, Burr RL, Cain KC, Newell DW, Mitchell PH. Effect of continuous display of cerebral perfusion pressure on outcomes in patients with traumatic brain injury. Am J Crit Care. 2006 Nov;15(6):600-9; quiz 610. PMID 17053267
- [Result] Kirkness CJ, Burr RL, Cain KC, Newell DW, Mitchell PH. Relationship of cerebral perfusion pressure levels to outcome in traumatic brain injury. Acta Neurochir Suppl. 2005;95:13-6. doi: 10.1007/3-211-32318-x_3. PMID 16463811
- [Result] Kirkness CJ, Burr RL, Thompson HJ, Mitchell PH. Temperature rhythm in aneurysmal subarachnoid hemorrhage. Neurocrit Care. 2008;8(3):380-90. doi: 10.1007/s12028-007-9034-y. PMID 18066502
- [Result] Thompson HJ, Kirkness CJ, Mitchell PH. Intensive care unit management of fever following traumatic brain injury. Intensive Crit Care Nurs. 2007 Apr;23(2):91-6. doi: 10.1016/j.iccn.2006.11.005. Epub 2007 Jan 12. PMID 17223560